CLINICAL TRIAL: NCT06054646
Title: Evaluation of Microinjected Amnion-derived Collagen by Dermapen in the Smoothing of Skin Wrinkles
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Egyptian Atomic Energy Authority (Other Government)
Collaborators: Waleed Nemr,Egyptian Atomic Energy Authority (Unknown)
Responsible Party: Principal Investigator, Nashwa Radwan, Head of amnion preparation laboratory, Egyptian Atomic Energy Authority
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3122019NCRRT
Record Dates: First submitted 2023-09-19; First posted 2023-09-26 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Facial Wrinkles - Rough Texture - Hyperpigmentation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amnion Collagen (Active Comparator): The right side of the split-face was treated by micro-injection of Amnion Collagen
  Interventions: Biological: Amnion collagen
- PRP (Active Comparator): The left side of the split-face was treated by micro-injection of Platelet-rich plasma (PRP)
  Interventions: Biological: Platelet-rich plasma

INTERVENTIONS:
Biological: Amnion collagen — A collagen extract sourced from the human amniotic membrane
  Arms: Amnion Collagen
Biological: Platelet-rich plasma — Autologous preparation of PRP
  Other Names: PRP
  Arms: PRP

SUMMARY:
The aim of this work was to assess the efficacy of irradiated amniotic collagen matrix in comparison with platelet rich plasma in facial rejuvenation.The present study included 20 patients with facial wrinkles divided into 2 groups using split face technique: Group (A) subjected to microneedling with amnion gel on the right side of the face . Group (B) subjected to microneedling with PRP on the other side of the face.According to a skin analysis camera (antera camera), there was statistically significant improvement after treatment and between both groups as regard to the roughness(texture) and melanin appeared by Antera camera in which group (A) showed better improvement than group (B). Also, skin biopsies showed improvement in both sides after treatment in which the epidermis was thicker, collagen bundles were broader and thicker than before treatment also elastic fibers were longer, evenly arranged and thicker than before treatment. The patients were followed up over a period of 3 months after the last session with no complications or changes were occurred and the results of sessions were maintained.

ELIGIBILITY:
Inclusion Criteria:

* Patients who did not receive any treatment for aging within the last 6 months.
* Patients who accepted to participate in this study.

Exclusion Criteria:

* Patients with bleeding, coagulation disorders, severe anemia, liver disease, renal disease, recurrent facial herpes, keloid formation, pregnant, and lactating females.

Ages: 36 Years to 57 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Because females are interested in facial rejuvenation more than males. So, this study targeted females.
Enrollment: 20 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-09-22 (Actual); Study Completion 2021-12-08 (Actual)

PRIMARY OUTCOMES:
Evaluation of facial wrinkles according to wrinkle severity rate scale (WSRS) | 2 weeks
  grade 0 = no wrinkles, grade I = just perceptible wrinkle, grade II = shallow wrinkles, grade III = moderately deep wrinkles, grade IV = deep wrinkle with well-defined edges, grade V = very deep wrinkle with redundant fold.
Evaluation of facial wrinkles according to Global Aesthetic Improvement Scale (GAIS) | 2 weeks
  No improvement or mild improvement less than 25% moderate improvement = 26%-50% marked improvement = 51%-75% excellent improvement = more than 75%
skin pigmentation assessed by skin hyper-pigmentation index | 2 weeks
  score: No pigmentation=1, sever pigmentation=4
Histopathology improvement of skin biopsy | 2 weeks
  improved skin structure=1, non-improved skin structure=0

CONTACTS AND LOCATIONS:
Locations (1):
- Egyptain Atomic Energy Authority, Cairo, Egypt